CLINICAL TRIAL: NCT00903825
Title: Optimization of Local Anesthetic Effect With Duplex Ultrasound Guided Injection of Lidocaine Before Femoral Artery Catheterization: A Prospective Randomized Controlled Trial
Brief Title: Duplex Guided Application of Local Anesthetic Before Femoral Artery Catheterization
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Siablis Dimitrios, Professor of Radiology, Patras University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44/27-2-09; 11/14.4.2009
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2009-05

CONDITIONS: Local Anesthetics; Ultrasound Guidance; Catheterization
Keywords: femoral artery puncture; local anesthesia; ultrasound guided
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual palpation (Active Comparator): Local anesthetic before femoral artery puncture will be injected with the classic manual palpation technique
  Interventions: Procedure: Injection of femoral local anesthetic (lidocaine) with manual palpation
- Ultrasound guidance (Experimental): Local anesthetic before femoral artery puncture will be performed with the use of duplex ultrasound guidance
  Interventions: Procedure: Ultrasound guided injection of femoral local anesthetic (lidocaine)

INTERVENTIONS:
Procedure: Ultrasound guided injection of femoral local anesthetic (lidocaine) — Injection of lidocaine (< 10 mls of lidocaine, 1%w/v) before femoral artery puncture with free-hand duplex ultrasound guidance.
  Arms: Ultrasound guidance
Procedure: Injection of femoral local anesthetic (lidocaine) with manual palpation — Injection of lidocaine before femoral artery catheterization with manual palpation.
  Arms: Manual palpation

SUMMARY:
The aim of this study is to evaluate the optimization of local anesthetic effect with duplex ultrasound-guided injection of lidocaine before femoral artery puncture during diagnostic or therapeutic interventional procedures.

In total, 200 patients scheduled for various diagnostic or therapeutic interventional radiology procedures requiring femoral artery puncture, will be randomized in two groups after informed consent. Patients will be randomized to undergo groin local anesthesia with the proposed method of duplex ultrasound guided injection of lidocaine versus standard injection of lidocaine with manual palpation (control group).

The protocol includes the registration of patients' demographics (age, gender, risk factors for peripheral arterial disease), arterial morphological characteristics (calcifications and presence of atheromatous disease), as well as technical details of the procedure (total puncture duration, sheath size, antegrade/retrograde puncture, etc.)

Primary study endpoint will be peri-procedural pain that will be assessed with the use of a visual analog scale (VAS) completed by the patient at the end of the procedure. Secondary study endpoints will evaluate procedural safety and complications during the immediate post-procedural period (up to 7 days).

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for diagnostic intra-arterial procedures
* Patient scheduled for therapeutic intra-arterial procedures
* At least 1 palpable femoral artery
* Patient informed consent

Exclusion Criteria:

* Allergic reaction to iodine contrast media
* Allergic reaction to lidocaine
* Bilateral obstruction of femoral arteries
* Impaired or lost vision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) for pain evaluation | immediatelly after sheath placement, days 0-7

SECONDARY OUTCOMES:
major and/or minor puncture site complications (infection, groin hematoma, pseudoaneurysm formation,arterio-venous fistula, major bleeding) | immediate, up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Siablis, Professor, Study Director — Department of Radiology, Patras University Hospital
Locations (1):
- Department of Radiology, Angiography Suite, Patras University Hospital, Pátrai, ACHAIA, Greece